CLINICAL TRIAL: NCT00343174
Title: Multicenter Parallel Randomized Double-Blind Placebo Controlled Study of Efficacy and Safety of Intravenous Ancrod ( Arvin ) Given Within 6 Hours After the Onset of Acute Ischemic Stroke: European Stroke Treatment With Ancrod Trial ESTAT
Brief Title: Intravenous Ancrod for the Treatment of Acute Ischemic Stroke Within 6 Hours After Onset of Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MPR-CC-0101
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2006-06-22 (Estimated); Status verified 2002-01

CONDITIONS: Brain Infarction; Cerebral Ischemia; Acute Stroke
Keywords: stroke; vascular diseases
MeSH Terms: conditions — Brain Infarction; Brain Ischemia; Stroke; Vascular Diseases | interventions — Ancrod

INTERVENTIONS:
Drug: Ancrod

SUMMARY:
Treatment of acute stroke is still difficult and the only specific drug approved (rtPA) can only be administered if treatment starts within 3 hours after onset of symptoms. This results in a still too small number of patients treated with rtPA ( < 15% in best clinical care institutions ). Ancrod is a differently acting biological drug which has been used for a long time but not for acute stroke treatment. STAT was the first RCT of medium size to show a significant benefit/risk ration if treatment starts within 3 hours. ESTAT was designed closely related to STAT but with a longer 6 hours window and specifically extended inclusion/exclusion criteria to avoid secondary complications possibly related to a longer time window.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above, both sexes
* Acute ischemic stroke with first symptoms within 6 hours of beginning
* Treatment after onset of symptoms
* SSS < 40 at baseline ( consciousness necessary )

Exclusion Criteria:

* Clinical or CT evidence of brain hemorrhage or hemorrhagic transformation
* CT evidence of major signs of developing infarction
* Coma
* Prior strokes within 6 weeks
* Severe hypertension (> 220 systolic > 120 mm Hg diastolic)
* Baseline fibrinogen < 100 mg/dL
* Recent use of thrombolytic agents
* Recent or anticipated surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: M G Hennerici, MD, Principal Investigator — Univ Heidelberg Klinikum Mannheim; Jean M Orgogozo, MD, Study Director — Univ Bordeaux France

REFERENCES:
- [Derived] Hennerici MG, Kay R, Bogousslavsky J, Lenzi GL, Verstraete M, Orgogozo JM; ESTAT investigators. Intravenous ancrod for acute ischaemic stroke in the European Stroke Treatment with Ancrod Trial: a randomised controlled trial. Lancet. 2006 Nov 25;368(9550):1871-8. doi: 10.1016/S0140-6736(06)69776-6. PMID 17126719